CLINICAL TRIAL: NCT07315100
Title: Image-guided Navigation During Robot-assisted Partial Nephrectomy
Brief Title: Navigated Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N24NPN
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Renal Cancer; Partial Nephrectomy
Keywords: Image Guided Surgery; Navigation; Robot-assisted partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: One group to evaluate the feasibility and accuracy of the proposed methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled for robot-assisted partial nephrectomy (Experimental): This study is designed as a single-center prospective feasibility study to evaluate the precision of EM tracking navigation in RAPN. We plan to conduct this study over a period of approximately 1 year. Eligible participants are patients who are scheduled for RAPN at the NKI-AvL, without restrictions on the pathology type of the lesions targeted for removal. Patients are informed about the study before the planned surgery and, after being provided with the necessary information regarding participation in the study, will be asked for informed consent. Participation in the study concludes at the end of the surgical procedure.
  Interventions: Procedure: Image guided surgery

INTERVENTIONS:
Procedure: Image guided surgery — Diagnostic CT and MRI scans are used to create a 3D digital model to illustrate the lesion's relation to the kidney and surrounding anatomy. The surgeon reviews this model, validates the segmentation, and plans the resection volume. The surgical procedure proceeds according to standard protocols in a standard operational setting, with the addition of navigation tools. A sterile EM sensor is inserted through a separate 5mm trocar and affixed to the kidney in proximity to the lesion in a region intended to be resected. Registration of the 3D model is conducted using an EM pointer or a tracked instrument, pointing to identifiable anatomical landmarks or structures on the kidney to validate accuracy. Both the digital model and the location of tracked instruments are displayed in real-time to the surgeon in the video console of the robot, allowing real-time navigation.

SUMMARY:
This study aims to evaluate electromagnetic (EM) tracked navigation in robot-assisted partial nephrectomy (RAPN), addressing kidney movement issues by attaching a tracked EM sensor close to the lesion. This assessment will be based on the navigation's ability to achieve preoperatively planned resection volumes aiming to assist in radical resection margins of the lesion. The current challenge for surgeons performing RAPN is to minimize the removal of healthy kidney tissue, as the rates of positive resections are very low. Additionally, the study aims to explore the practical application of image guidance in RAPN, evaluating aspects such as duration, surgical and technical success, and the surgeons' perceptions. Ultimately, this research seeks to determine if the addition of navigation can enhance RAPN outcomes, particularly in terms of kidney tissue preservation and radical lesion removal. The success of this technique could result in broader adoption of kidney-sparing surgeries, even in complex scenarios where radical resection is at risk.

DETAILED DESCRIPTION:
Robot-assisted partial nephrectomy (RAPN) is now the preferred option for treatable renal lesions due to its ability to preserve kidney function while effectively treating cancer. Despite RAPN's effectiveness, its surgical complexity and varied approach requirements pose challenges. Image-guided surgery applies pre-operative imaging for patient-specific intra-operative visualization of the kidney and lesion margins to support the surgeon during resection. However, adapting to surgery-induced deformations remains a challenge. An approach that is able to correct for organ movements during surgery might result in an optimal preservation rate of healthy kidney parenchyma and improved decisiveness for the surgeon during resection. On the long term, this might result in a larger shift from radical to partial nephrectomies, leading to patients with improved renal functions after lesion resection.

The primary objective is to assess the ability to achieve preoperatively planned resection volumes by adding EM tracked navigation in RAPN, as minimizing the removal of healthy kidney tissue is challenging nowadays. A deviation within 35% between the planned and actual resection volumes is considered comparable and therefore deemed successful. Secondary objectives are the time for localizing and removing the renal lesion, the impact on surgical decisiveness, and the clinical and technical success of implementing the navigation setup.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient provides written informed consent form
* Patient is scheduled for robot-assisted partial nephrectomy

Exclusion Criteria:

* Ferro-magnetic implants or other factors in the abdominal or thoracic area that could influence image quality
* Pacemaker or defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Accuracy of the EM navigation setup in preserving the volume of renal tissue designated for resection prior to surgery | One day
  The planned resection volume will be compared to the actual resected volume using CT scan data. A navigation is deemed successful if comparable resection volumes are measured. The criteria for comparable resection volume measurement is defined as a discrepancy of no more than 35% between the preoperative and post-operative volumes, ensuring that the navigation aids in achieving precision in surgical outcomes. The study is successful when 70% of the navigations (i.e. 14 out of 20 patients) are successful.

SECONDARY OUTCOMES:
Time required for navigation implementation | One day
Clinical success of number of negative resection margins | One day
Technical usability of the navigation setup using post-operative questionnaires for surgeons | One day

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided